CLINICAL TRIAL: NCT02150265
Title: Effectiveness of Cognitive Behavioral Short-term Treatment for Adolescents With Emotional Symptom Problems in Community Clinics in Norway. A Randomized Controlled Study
Brief Title: Effectiveness of Six Sessions CBT for Adolescents With Emotional Problems in Community Clinics
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: The Royal Norwegian Ministry of Health (Other); Regionsenter for barn og unges psykiske helse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/1937; 8563/PFP1112-13 (Other Grant/Funding Number: Northern Norway Regional Health Authority (Helse Nord RHF))
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Generalized Anxiety Disorder; Social Phobia; Agoraphobia; Depression; Panic Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Agoraphobia; Depression; Panic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting list control group (No Intervention): 6 week waiting list
- Individual cognitive behavioral therapy with SMART (Experimental): SMART manual cognitive behavioral therapy individual weekly sessions for 6 weeks
  Interventions: Behavioral: SMART manual cognitive behavioral therapy

INTERVENTIONS:
Behavioral: SMART manual cognitive behavioral therapy
  Arms: Individual cognitive behavioral therapy with SMART

SUMMARY:
Background: There is need for more effectiveness studies concerning treatment of emotional symptom problems indicating anxiety and depression in adolescents. SMART is the only treatment manual for combined emotional disorders developed in Norwegian.

Purpose: To find the best individualized treatment for adolescents with emotional difficulties by: Finding criteria for the selection of appropriate patients for treatment with cognitive-behavior therapy program SMART in an outpatient population (14-18 years). Finding predictors of completion of treatment program SMART. Examining the effects of treatment with the SMART program at 6 months follow-up.

Design: A randomized controlled study in six outpatient clinics in the north of Norway. N= 160 referred adolescents (14-18 years) with score above 6 on the Emotional Problems scale of the Strength and Difficulties Questionnaire (SDQ). Two thirds are treated according to the SMART-manual immediately, while the waiting list control group is treated with SMART after six weeks.

Hypothesis: The SMART treatment is an effective treatment for emotional symptom problems.

Publication: The results sought published internationally and nationally and will be communicated to clinicians.

ELIGIBILITY:
Inclusion Criteria:

Age 14 to 18 years Referred to Community Mental Health Clinic for Children and Adolescents

* Score above 6 on Emotional symptoms scale on the SDQ Fluent Norwegian language

Exclusion Criteria:

* Indicators for Pervasive Developmental Disorder (PDD) Acute suicidal symptoms Psycho-active drug treatment start coinciding with start of intervention Symptoms indicating psychotic disorder

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 163 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Status of primary emotional disorder based on theDevelopment and Well-Being Assessment (DAWBA) interview schedule with parents and youths | At recruitment, before treatment start and at 6 months follow up
  Diagnostic interview

SECONDARY OUTCOMES:
SDQ Strengths and Difficulties Questionnaire | At recruitment, before treatment start and at 6 months follow up
  Measure of general emotional and behavioral symptoms and strengths
Anxiety symptom score on the Multi-Dimensional Anxiety Scale for Children (MASC) | At recruitment, before treatment start and at 6 months follow up
  Measure of anxiety symptoms
Depression symptom status as measured by the self-rating instrument Beck Depression Inventory (BDI-II) | At recruitment, before treatment start and at 6 months follow up
  Measure of depressive symptoms
Life functioning as measured by the rating scale C-GAS rated by clinicians | At recruitment, before treatment start and at 6 months follow up
  Measure of functioning
General outcome measured by Clinical Outcomes in Routine Evaluations Outcome Measure (CORE-OM) | At recruitment, before treatment start and at 6 months follow up. The short version (CORE 10) mid-therapy: 3 weeks after starting treatment
  Measure of symptoms, risk, functioning and total burden of disorder

CONTACTS AND LOCATIONS:
Overall Officials: Ingunn Skre, PhD, Principal Investigator — UiT Arctic University of Norway; Simon-Peter Neumer, Dr philos, Study Chair — Regionsenter for barn og unges psykiske helse, Sør-Øst
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Lorentzen V, Fagermo K, Handegard BH, Neumer SP, Skre I. Long-term effectiveness and trajectories of change after treatment with SMART, a transdiagnostic CBT for adolescents with emotional problems. BMC Psychol. 2022 Jul 5;10(1):167. doi: 10.1186/s40359-022-00872-y. PMID 35791020
- [Derived] Lorentzen V, Fagermo K, Handegard BH, Skre I, Neumer SP. A randomized controlled trial of a six-session cognitive behavioral treatment of emotional disorders in adolescents 14-17 years old in child and adolescent mental health services (CAMHS). BMC Psychol. 2020 Mar 14;8(1):25. doi: 10.1186/s40359-020-0393-x. PMID 32171328